CLINICAL TRIAL: NCT06656260
Title: Validation of Ocular Pain Questionnaire: Single-center, Prospective Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Giulio Ferrari, Professor of Ophthalmology-San Raffaele Vita Salute University, Cornea and Ocular Surface Unit; Head-Eye Repair Lab San Raffaele Scientific Institute, IRCCS Ospedale San Raffaele
Other Study IDs: QDO
Record Dates: First submitted 2024-07-30; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Ocular Pain; OSDI; OPAS
Keywords: Ocular pain; OSDI; OPAS; Questionnaire
MeSH Terms: conditions — Eye Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study will be a single-center, observational, prospective validation study with survey and sample characteristics comparable to similar validation studies in the literature.

Pain represents a physiological response to the presence of tissue damage and is associated with numerous pathological conditions of the ocular surface.

Furthermore, in the presence of dysfunction of the nociceptive system, ocular pain can occur chronically with neuropathic features.

Pain quantification systems used to guide symptomatic therapy include the Ocular Surface Disease Index (OSDI); the Ocular Pain Assessment Survey (OPAS); and the Standardized Patient Evaluation of Eye Dryness (SPEED).

The OSDI assesses the presence of ocular symptoms, their impact on activities of daily living, and the presence of any aggravating factors. Although it is used in clinical practice and research activities in a translated version, it has never been validated in Italian.

The OPAS studies in more detail the characteristics of pain and associated symptoms and their impact on the patient's overall quality of life. This instrument has neither been translated nor validated in an Italian version.

The failure to validate the OSDI and OPAS questionnaires in the Italian version marks the starting point for this validative study.

The SPEED questionnaire, already translated and validated in Italian, will be used as the Gold Standard and will allow comparison of the other instruments.

Finally, six questions regarding imaginary scenarios of pain experiences will be proposed to assess the individual threshold of nociceptive sensitivity taken from the Pain Sensitivity Questionnaire (two for mild pain assessment, two for intermediate intensity stimuli, and two for intense pain situations).

Therefore, the primary objective of the study is to validate the Italian version of the OSDI and OPAS questionnaires while the secondary objective is to analyze the responses to the questionnaires by subgroups of general sensitivity to nociceptive stimuli.

ELIGIBILITY:
Inclusion Criteria:

* NA

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of patients with corneal and ocular surface diseases referred to the Ophthalmology O.U. - Cornea Center of IRCCS Ospedale San Raffaele will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 333 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study is to validate the Italian version of the OSDI and OPAS questionnaires. | The questionnaire will be acquired at day 0 (first time-point) and at day 7 (second time-point)

SECONDARY OUTCOMES:
Secondary objective is the analysis of questionnaire responses by subgroups of general sensitivity to nociceptive stimuli. | The questionnaire will be acquired at day 0 (first time-point) and at day 7 (second time-point)